CLINICAL TRIAL: NCT03464578
Title: Evidence Based Algorithm to Treat Patients With Proximal Humerus Fractures - A Prospective Study With Early Clinical and Overall Performance Results
Brief Title: Evidence Based Algorithm for Proximal Humerus Fractures
Status: Completed | Type: Observational
Sponsor: Cantonal Hospital of St. Gallen (Other)
Responsible Party: Principal Investigator, Bernhard Jost, Prof. Dr. med, Head of Departement, Cantonal Hospital of St. Gallen
Other Study IDs: ProxHumFx
Record Dates: First submitted 2018-03-01; First posted 2018-03-14 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Proximal Humeral Fracture
MeSH Terms: conditions — Shoulder Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Therapy of proximal humeral fractures (irrespective conservative or operative)

SUMMARY:
Proximal humerus fractures are particularly frequent injuries and represent 6% of all fractures with an overall incidence of 63/100.000 in human. The goal is to assess our institutional evidence based algorithm for treatment of proximal humeral fractures.

Objective(s):

1. Test the algorithm in terms of clinical applicability and clinical outcome
2. Compare general outcome and general complication/revision rate to the literature.

Inclusion / Exclusion criteria: Inclusion: All patients with an acute proximal humeral fracture (not older than 48 hours) admitted to our institution later than 1.1.2014. Exclusion: Multilevel and pathological fractures are excluded.

Terminally ill patients and those not being able, or willing to sing the informed consent.

Project Centre(s): Single-centre.

Statistical Considerations: Standard descriptive statistics will be performed using R-statistics program. Considering the population of 160 patients, we will be able to detect differences in proportions as low as 0.15 with power 82% and alpha = 0.05.

Other methodological Considerations: Terms applicability of a treatment protocol and adhesion to protocol are not well defined for decision making in orthopaedic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Acute traumatic proximal humeral fracture
* Signed informed consent

Exclusion Criteria:

* Fracture older than 48 hours at admission
* Multilevel fractures of the humerus
* Pathological fractures
* Terminally ill patients.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with an acute proximal humeral fracture admitted to our institution.
Sampling Method: Non-Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Constant Score | One year
  Point 0-100

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Jost, MD, Study Director — Head of the departement
Locations (1):
- Department of Orthopaedic Surgery and Traumatology, Sankt Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: No